CLINICAL TRIAL: NCT04237532
Title: Effectiveness of Sublingual Versus Intranasal Administration of Dexmedetomidine for Sedation of Children Undergoing Dental Treatment (A Randomized Controlled Clinical Trial)
Brief Title: Sublingual Versus Intranasal Administration of Dexmedetomidine for Sedation of Children Undergoing Dental Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health; Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sublingual vs intranasal DEX
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Anti-anxiety Agents; Moderate Sedation

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled clinical trial with a cross over design where each patient will serve as his/her own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Dexmedetomidine (Experimental)
  Interventions: Drug: Intranasal Dexmedetomidine
- Sublingual Dexmedetomidine (Experimental)
  Interventions: Drug: Sublingual Dexmedetomidine

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine — The mucosal atomizing device will be used intranasally where the sedative drug will be equally divided and sprayed into each nostril while the child semi reclined position.
  Arms: Intranasal Dexmedetomidine
Drug: Sublingual Dexmedetomidine — The mucosal atomizing device will be used sublingually by asking the child to touch their maxillary incisor teeth with the tip of their tongue and instruct the child not to swallow the drug for 30 seconds.
  Arms: Sublingual Dexmedetomidine

SUMMARY:
The aim of this study is to assess the efficacy of Dexmedetomidine drug either used sublingually or intranasally in managing healthy children during dental treatment

DETAILED DESCRIPTION:
Each child should fulfill the requirements of having a dental condition which needs treatment in two dental sessions, where each session should not exceed thirty minutes. At the first visit ,either sublingual or intranasal Dexmedetomidine will be used, while at the second visit the alternate route will be implemented in a cross-over design. At least one week interval between the two visits will be secured.

ELIGIBILITY:
Inclusion Criteria:

* Frankl behavior rating score 2.
* ASA I physical status.
* Dental intervention under local anesthesia not requiring more than 30 minutes.
* No previous dental experience.
* Parent/guardian written consent.

Exclusion Criteria:

* Dental treatment indicated requiring general anesthesia.
* Mouth breathers.
* Patients with acute upper respiratory illness.
* Medically compromised patients.
* Cognitively impaired patients.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Acceptance of drug administration | during the sedation procedure
  Assessed by a 4 point Likert scale as follows: 1 (Good) the child accepted the drug without any refusal. 2 (fair) the child accepted the drug with some verbal resistance. 3 (poor) the child accepted the drug with some physical resistance. 4 (refused) the child refused but drug administration was possible after persuation.
Level of Sedation | during the sedation procedure
  Time taken by both routes to reach the desired level of sedation using Wilton et al sedation scale and it is scored as follows: 1. Agitated: Clinging parent and/or crying. 2.Alert: Awake, but not clinging to parent may whimper but not crying. 3.Calm: Sitting or lying comfortably with eyes spontaneously open. 4.Drowsy: Sitting or lying comfortably with eyes spontaneously closing but responds to minor stimulation. 5. Asleep: Eyes closed, rousable, does not respond to minor stimulation.
Anxiety level | during the sedation procedure
  Anxiety level during local anesthesia administration will be evaluated using Venham's clinical anxiety scale. 0: Relaxed child, 1: Uneasy, concerned, 2:Child appears scared, 3:Shows reluctance to enter situation, difficulty in correctly assessing situational threat, 4:Anxiety interferes with ability to assess situation.

CONTACTS AND LOCATIONS:
Overall Officials: May Shaat, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Niveen Bakry, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Dalia M Talaat, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Ahmed M El-Shafei, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] al-Rakaf H, Bello LL, Turkustani A, Adenubi JO. Intra-nasal midazolam in conscious sedation of young paediatric dental patients. Int J Paediatr Dent. 2001 Jan;11(1):33-40. doi: 10.1046/j.1365-263x.2001.00237.x. PMID 11309871
- [Background] Wilton NC, Leigh J, Rosen DR, Pandit UA. Preanesthetic sedation of preschool children using intranasal midazolam. Anesthesiology. 1988 Dec;69(6):972-5. doi: 10.1097/00000542-198812000-00032. No abstract available. PMID 3195771
- [Background] Venham LL, Gaulin-Kremer E, Munster E, Bengston-Audia D, Cohan J. Interval rating scales for children's dental anxiety and uncooperative behavior. Pediatr Dent. 1980 Sep;2(3):195-202. No abstract available. PMID 6938934